CLINICAL TRIAL: NCT00405236
Title: A Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Changes in Inflammatory Markers in Induced Sputum Following Treatment With Tiotropium Inhalation Capsules 18mcg Once Daily in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Tiotropium on Inflammation and Exacerbations in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Free and University College Medical School (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.270
Record Dates: First submitted 2006-11-27; First posted 2006-11-29 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: inflammation; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium

SUMMARY:
Patients with COPD experience exacerbations that are a major cause of morbidity. Exacerbations are associated with increased airway and systemic inflammation and those experiencing frequent exacerbations demonstrate increased inflammation in the stable state. Tiotropium has been shown to reduce exacerbation frequency and it might be postulated that this is due to a reduction in inflammation. The study will compare airway inflammation and exacerbation frequency in patients with COPD on tiotropium or placebo.

DETAILED DESCRIPTION:
Patients with COPD will be randomised to tiotropium or placebo in addition to their usual medication. They will be followed prospectively over 1 year and provide sputum for quantification of IL-6 and IL-8 at baseline and at 3 monthly intervals.Serum IL-6 will also be quantified at baseline and over the year. Changes in inflammatory markers will be assessed by analysis of area under the curve of log transformed data. Exacerbation frequency will be calculated from patient diary cards using a previously validated symptom-based exacerbation definition.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of COPD,
* FEV1 < 80% predicted,
* minimum 10 pack year smoking history

Exclusion Criteria:

* asthma,
* atopic disease,
* eosinophilia,
* history of malignancy,
* history of clinically significant pulmonary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220
Dates: Start 2002-10; Study Completion 2005-01

PRIMARY OUTCOMES:
sputum IL-6

SECONDARY OUTCOMES:
sputum IL-8
sputum MPO
serum IL-6
serum CRP
exacerbation frequency
FEV1
FVC

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga A Wedzicha, MD, Principal Investigator — Academic Unit of Respiratory Medicine, Royal Free and University College Medical School
Locations (1):
- London Chest Hospital, London, United Kingdom